CLINICAL TRIAL: NCT02809183
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Efficacy of TRC101 in Subjects With Chronic Kidney Disease and Low Serum Bicarbonate Levels
Brief Title: Evaluation of TRC101 in Subjects With Chronic Kidney Disease and Metabolic Acidosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tricida, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRCA-101; 2015-004327-31 (EudraCT Number)
Record Dates: First submitted 2016-06-14; First posted 2016-06-22 (Estimated); Results first posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Acidosis
Keywords: metabolic acidosis; serum bicarbonate; kidney disease
MeSH Terms: conditions — Acidosis; Kidney Diseases | interventions — veverimer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo-BID (Placebo Comparator): Administered twice daily (BID) for 14 days
  Interventions: Drug: Placebo
- TRC101 (1.5g BID) (Experimental): Administered twice daily (BID) for 14 days
  Interventions: Drug: TRC101
- TRC101 (3g BID) (Experimental): Administered twice daily (BID) for 14 days
  Interventions: Drug: TRC101
- TRC101 (4.5g BID) (Experimental): Administered twice daily (BID) for 14 days
  Interventions: Drug: TRC101
- TRC101 (6g QD) (Experimental): Administered once daily (QD) for 14 days
  Interventions: Drug: TRC101
- Placebo-QD (Placebo Comparator): Administered once daily (QD) for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — oral suspension
  Arms: Placebo-BID; Placebo-QD
Drug: TRC101 — oral suspension
  Other Names: Veverimer
  Arms: TRC101 (1.5g BID); TRC101 (3g BID); TRC101 (4.5g BID); TRC101 (6g QD)

SUMMARY:
This was a double-blind, placebo-controlled, parallel-design, 6-arm, fixed dose study. The study enrolled 135 adult male and female subjects with Stage 3 or 4 chronic kidney disease and low serum bicarbonate levels. The study was conducted in two parts. In Part 1 study drug dosing (TRC101 or placebo) continued for 14 days twice daily (BID). In Part 2 study drug dosing (TRC101 or placebo) continued for 14 days once daily (QD).

The maximum study duration per subject was anticipated to be up to 42 days.

ELIGIBILITY:
Inclusion Criteria:

* Estimated glomerular filtration rate (eGFR) of 20 to <60 mL/min/1.73m2
* Serum bicarbonate level of 12 to 20 mEq/L

Exclusion Criteria:

* Any level of low serum bicarbonate that, in the opinion of the Investigator, requires emergency intervention.
* Severe comorbid conditions other than chronic kidney disease.
* Chronic obstructive pulmonary disease.
* Anticipated changes in doses of any of the following drugs or drug classes: diuretics, non-ophthalmic carbonic anhydrase inhibitors, oral diabetes drugs, antihypertensive drugs, antacids, H2-blockers, or proton pump inhibitors.
* Excluded drugs or drug classes: insulin, non-daily or "as needed" diuretics, herbal products, dietary supplements, multivitamins, naturopathic remedies, sodium bicarbonate, potassium citrate, sodium citrate or other alkali therapy, non-steroidal anti-inflammatory drugs (NSAIDs), fiber supplements, laxatives, calcium and magnesium supplements, or electrolyte binders and other binder drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Stasiv, PhD, Study Director — Tricida, Inc.
Locations (5):
- Investigative Site 1, Sofia, Bulgaria
- Georgia (4):
  - Investigative Site 3, Tbilisi
  - Investigative Site 4, Tbilisi
  - Investigative Site 5, Tbilisi
  - Investigative Site 6, Tbilisi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bushinsky DA, Hostetter T, Klaerner G, Stasiv Y, Lockey C, McNulty S, Lee A, Parsell D, Mathur V, Li E, Buysse J, Alpern R. Randomized, Controlled Trial of TRC101 to Increase Serum Bicarbonate in Patients with CKD. Clin J Am Soc Nephrol. 2018 Jan 6;13(1):26-35. doi: 10.2215/CJN.07300717. Epub 2017 Nov 4. PMID 29102959

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo BID: Placebo administered twice daily (BID) for 14 days
- 1.5g TRC101 BID: 1.5g TRC101 administered twice daily (BID) for 14 days
- 3g TRC101 BID: 3g TRC101 administered twice daily (BID) for 14 days
- 4.5g TRC101 BID: 4.5g TRC101 administered twice daily (BID) for 14 days
- Placebo QD: Placebo administered once daily (QD) for 14 days
- 6g TRC101 QD: 6g TRC101 administered once daily (QD) for 14 days
Period: Overall Study
Arm/Group | Placebo BID | 1.5g TRC101 BID | 3g TRC101 BID | 4.5g TRC101 BID | Placebo QD | 6g TRC101 QD
Started | 25 | 25 | 25 | 26 | 6 | 28
Completed | 25 | 25 | 25 | 26 | 6 | 28
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population
Groups:
- Pooled Placebo: Pooled placebo treatment groups (Placebo administered twice daily [BID] for 14 days + Placebo administered once daily [QD] for 14 days)
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | 1.5g TRC101 BID | 3g TRC101 BID | 4.5g TRC101 BID | 6g TRC101 QD | Total
Number analyzed (Participants) | 31 | 25 | 25 | 26 | 28 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (12) | 58 (14) | 60 (13) | 61 (13) | 63 (11) | 60.3 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 8 | 11 | 12 | 49
  Male | 19 | 19 | 17 | 15 | 16 | 86
Diabetes [Count of Participants; unit: Participants] | 20 | 18 | 20 | 19 | 17 | 94
Hypertension [Count of Participants; unit: Participants] | 30 | 24 | 23 | 23 | 26 | 126
Heart Failure [Count of Participants; unit: Participants] | 7 | 5 | 7 | 5 | 5 | 29
Serum Bicarbonate [Mean (Standard Deviation); unit: mEq/L] | 17.6 (1.4) | 18.0 (1.0) | 17.8 (1.2) | 17.5 (1.3) | 17.7 (1.0) | 17.72 (1.197)
eGFR [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 34 (14) | 35 (13) | 40 (13) | 35 (13) | 31 (10) | 35.70 (12.419)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs) and Number of Subjects Who Discontinued Study Drug Due to a TEAE
Description: The number and percentage of subjects who reported treatment-emergent adverse events (TEAEs) summarized by system organ class and preferred term (see Reported Adverse Events) as well as by severity, causality, seriousness, and action taken with regard to study drug. All analyses were descriptive.
Time Frame: Through treatment period completion (Day 15)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | 1.5g TRC101 BID | 3g TRC101 BID | 4.5g TRC101 BID | 6g TRC101 QD
Number analyzed (Participants) | 31 | 25 | 25 | 26 | 28
Participants
  Subjects Reporting any TEAE | 14 | 13 | 9 | 17 | 17
  ≥ 1 Mild TEAE | 11 | 9 | 8 | 14 | 15
  ≥ 1 Moderate TEAE | 3 | 4 | 1 | 3 | 2
  ≥ 1 Severe TEAE | 0 | 0 | 0 | 0 | 0
  ≥ 1 Serious TEAE | 0 | 0 | 0 | 0 | 0
  Study Drug Discontinuation Due to TEAE | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Change From Baseline to the End of Treatment (Day 15) in Serum Bicarbonate Within Each Individual TRC101 Dose Group
Description: Serum bicarbonate at Day 15 minus serum bicarbonate at Baseline
Time Frame: Baseline and Day 15
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Arm/Group | Pooled Placebo | 1.5g TRC101 BID | 3g TRC101 BID | 4.5g TRC101 BID
Number analyzed (Participants) | 31 | 25 | 25 | 26
mEq/L | -0.2 (0.4) | 3.2 (0.4) | 3.0 (0.4) | 3.7 (0.4)
Statistical Analysis 1: Comparison: Pooled Placebo; Test type: Other — Single-group test; p = 0.5547, Mixed Models Analysis — The null hypothesis is that the mean change from baseline within the Pooled Placebo treatment group = 0 mEq/L; Group LS mean = -0.2, 95% CI 2-sided [-0.9 to 0.5], Standard Error of Mean 0.4
Statistical Analysis 2: Comparison: 1.5g TRC101 BID; The null hypothesis is that the mean change from baseline within the 1.5g TRC101 BID treatment group = 0 mEq/L; Test type: Other — Single-group test; p < 0.0001, Mixed Models Analysis — The null hypothesis is that the mean change from baseline within the 1.5g TRC101 BID group = 0 mEq/L; Group LS mean = 3.2, 95% CI 2-sided [2.4 to 4.0], Standard Error of Mean 0.4
Statistical Analysis 3: Comparison: 3g TRC101 BID; Test type: Other — Single-group test; p < 0.0001, Mixed Models Analysis — The null hypothesis is the 3g TRC101 BID treatment group mean change from baseline = 0 mEq/L; Group LS mean = 3.0, 95% CI 2-sided [2.2 to 3.8], Standard Error of Mean 0.4
Statistical Analysis 4: Comparison: 4.5g TRC101 BID; Test type: Other — Single-group test; p < 0.0001, Mixed Models Analysis — The null hypothesis is the 4.5g TRC101 BID treatment group mean change from baseline = 0 mEq/L; Group LS mean = 3.7, 95% CI 2-sided [2.9 to 4.5], Standard Error of Mean 0.4

3. Secondary Outcome: Comparison of Change From Baseline in Serum Bicarbonate at Day 15 Between Each TRC101 Dose Group Versus Placebo
Description: Serum bicarbonate at Day 15 minus serum bicarbonate at Baseline for each TRC101 dose group versus that for Placebo
Time Frame: Baseline and Day 15
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Arm/Group | Pooled Placebo | 1.5g TRC101 BID | 3g TRC101 BID | 4.5g TRC101 BID
Number analyzed (Participants) | 31 | 25 | 25 | 26
mEq/L | -0.2 (0.4) | 3.2 (0.4) | 3.0 (0.4) | 3.7 (0.4)
Statistical Analysis 1: Comparison: Pooled Placebo vs 1.5g TRC101 BID; Test type: Other — Two-group test; p < 0.0001, Mixed Models Analysis — The null hypothesis is the difference between treatment groups (1.5g TRC101 BID - Pooled Placebo) in the mean change from baseline = 0 mEq/L; Difference between group LS means = 3.4, 95% CI 2-sided [2.3 to 4.5], Standard Error of Mean 0.5
Statistical Analysis 2: Comparison: Pooled Placebo vs 3g TRC101 BID; Test type: Other — Two-group test; p < 0.0001, Mixed Models Analysis — The null hypothesis is the difference between treatment groups (3g TRC101 BID - Pooled Placebo) in the mean change from baseline = 0 mEq/L; Difference between group LS means = 3.2, 95% CI 2-sided [2.2 to 4.3], Standard Error of Mean 0.5
Statistical Analysis 3: Comparison: Pooled Placebo vs 4.5g TRC101 BID; Test type: Other — Two-group test; p < 0.0001, Mixed Models Analysis — The null hypothesis is the difference between the treatment groups (4.5g TRC101 BID - Pooled Placebo) in the mean change from baseline = 0 mEq/L; Difference between group LS means = 3.9, 95% CI 2-sided [2.9 to 5.0], Standard Error of Mean 0.5

4. Secondary Outcome: Change From Baseline in Serum Bicarbonate at Day 15 Within the Combined TRC101 Treatment Group
Description: Serum bicarbonate at Day 15 minus serum bicarbonate at Baseline
Time Frame: Baseline and Day 15
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Groups:
- Combined TRC101: Combined groups treated with TRC101 for 14 days (TRC101 BID: 1.5g, 3g and 4.5g; TRC101 QD: 6g)
Arm/Group | Combined TRC101
Number analyzed (Participants) | 104
mEq/L | 3.3 (0.2)
Statistical Analysis 1: Comparison: Combined TRC101; Test type: Other — Single-group test; p < 0.0001, Mixed Models Analysis — The null hypothesis is that the mean change from baseline within the Combined TRC101 treatment group = 0 mEq/L; Group LS mean = 3.3, 95% CI 2-sided [3.0 to 3.7], Standard Error of Mean 0.2

5. Secondary Outcome: Comparison of Change From Baseline in Serum Bicarbonate at Day 15 Between the Combined TRC101 Treatment Group Versus Placebo
Description: Serum bicarbonate at Day 15 minus serum bicarbonate at Baseline for the Combined TRC101 Treatment Group versus that for Placebo
Time Frame: Baseline and Day 15
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Arm/Group | Pooled Placebo | Combined TRC101
Number analyzed (Participants) | 31 | 104
mEq/L | -0.2 (0.4) | 3.3 (0.2)
Statistical Analysis 1: Comparison: Pooled Placebo vs Combined TRC101; Test type: Other — Two-group test; p < 0.0001, Mixed Models Analysis — The null hypothesis is that the difference between treatment groups (Combined TRC101 - Pooled Placebo) in the mean change from baseline = 0 mEq/L; Difference between group LS means = 3.6, 95% CI 2-sided [2.8 to 4.4], Standard Error of Mean 0.4

6. Secondary Outcome: Comparison of the Proportion of Subjects Whose Serum Bicarbonate Values Increased From Baseline to Day 15 by Greater Than or Equal to 2, 3, or 4 mEq/L Between Each TRC101 Dose Group Versus Placebo
Description: Comparison of the proportion of subjects whose serum bicarbonate values increased from Baseline to Day 15 by greater than or equal to 2, 3, or 4 mEq/L between each TRC101 BID Dose Group versus Placebo
Time Frame: Baseline and Day 15
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | 1.5g TRC101 BID | 3g TRC101 BID | 4.5g TRC101 BID
Number analyzed (Participants) | 31 | 25 | 25 | 26
Participants
  => 2 mEq/L Baseline Serum Bicarbonate | 4 | 18 | 14 | 19
  => 3 mEq/L Baseline Serum Bicarbonate | 2 | 14 | 10 | 16
  => 4 mEq/L Baseline Serum Bicarbonate | 1 | 8 | 10 | 11
Statistical Analysis 1: Comparison: Pooled Placebo vs 1.5g TRC101 BID; Test type: Other — Two-group test; p < 0.0001, Fisher Exact — The null hypothesis is that the difference between treatment groups (1.5g TRC101 BID - Pooled Placebo) in proportion of subjects whose serum bicarbonate increased from baseline to Day 15 by => 2 mEq/L = 0
Statistical Analysis 2: Comparison: Pooled Placebo vs 1.5g TRC101 BID; Test type: Other — Two-group test; p < 0.0001, Fisher Exact — The null hypothesis is that the difference between treatment groups (1.5g TRC101 BID - Pooled Placebo) in proportion of subjects whose serum bicarbonate increased from baseline to Day 15 by => 3 mEq/L = 0
Statistical Analysis 3: Comparison: Pooled Placebo vs 1.5g TRC101 BID; Test type: Other — Two-group test; p = 0.0074, Fisher Exact — The null hypothesis is that the difference between treatment groups (1.5g TRC101 BID - Pooled Placebo) in proportion of subjects whose serum bicarbonate increased from baseline to Day 15 by => 4 mEq/L = 0
Statistical Analysis 4: Comparison: Pooled Placebo vs 3g TRC101 BID; Test type: Other — Two-group test; p = 0.0012, Fisher Exact — The null hypothesis is that the difference between treatment groups (3g TRC101 BID - Pooled Placebo) in proportion of subjects whose serum bicarbonate increased from baseline to Day 15 by => 2 mEq/L = 0
Statistical Analysis 5: Comparison: Pooled Placebo vs 3g TRC101 BID; Test type: Other — Two-group test; p = 0.0032, Fisher Exact — The null hypothesis is that the difference between treatment groups (3g TRC101 BID - Pooled Placebo) in proportion of subjects whose serum bicarbonate increased from baseline to Day 15 by => 3 mEq/L = 0
Statistical Analysis 6: Comparison: Pooled Placebo vs 3g TRC101 BID; Test type: Other — Two-group test; p = 0.0013, Fisher Exact — The null hypothesis is that the difference between treatment groups (3g TRC101 BID - Pooled Placebo) in proportion of subjects whose serum bicarbonate increased from baseline to Day 15 by => 4 mEq/L = 0
Statistical Analysis 7: Comparison: Pooled Placebo vs 4.5g TRC101 BID; Test type: Other — Two-group test; p < 0.0001, Fisher Exact — The null hypothesis is that the difference between treatment groups (4.5g TRC101 BID - Pooled Placebo) in proportion of subjects whose serum bicarbonate increased from baseline to Day 15 by => 2 mEq/L = 0
Statistical Analysis 8: Comparison: Pooled Placebo vs 4.5g TRC101 BID; Test type: Other — Two-group test; p < 0.0001, Fisher Exact — The null hypothesis is that the difference between treatment groups (4.5g TRC101 BID - Pooled Placebo) in proportion of subjects whose serum bicarbonate increased from baseline to Day 15 by => 3 mEq/L = 0
Statistical Analysis 9: Comparison: Pooled Placebo vs 4.5g TRC101 BID; Test type: Other — Two-group test; p < 0.0006, Fisher Exact — The null hypothesis is that the difference between treatment groups (4.5g TRC101 BID - Pooled Placebo) in proportion of subjects whose serum bicarbonate increased from baseline to Day 15 by => 4 mEq/L = 0

7. Secondary Outcome: Change From Baseline in Serum Bicarbonate at Day 15 Within the TRC101 6g QD Dose Group
Description: Serum bicarbonate at Day 15 minus serum bicarbonate at Baseline
Time Frame: Baseline and Day 15
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Arm/Group | 6g TRC101 QD
Number analyzed (Participants) | 28
mEq/L | 3.5 (0.4)
Statistical Analysis 1: Comparison: 6g TRC101 QD; Test type: Other — Single-group test; p < 0.0001, Mixed Models Analysis — The null hypothesis is that the mean change from baseline within the 6g TRC101 QD group = 0 mEq/L; Group LS mean = 3.5, 95% CI 2-sided [2.7 to 4.2], Standard Error of Mean 0.4

8. Secondary Outcome: Change From Baseline in Serum Bicarbonate at Day 15 Comparison Between the TRC101 6g QD Dose Group Versus Placebo
Description: Serum bicarbonate at Day 15 minus serum bicarbonate at Baseline for the TRC101 6g dose group versus that for Placebo
Time Frame: Baseline and Day 15
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Arm/Group | Pooled Placebo | 6g TRC101 QD
Number analyzed (Participants) | 31 | 28
mEq/L | -0.2 (0.4) | 3.5 (0.4)
Statistical Analysis 1: Comparison: Pooled Placebo vs 6g TRC101 QD; Test type: Other — Two-group test; p < 0.0001, Mixed Models Analysis — The null hypothesis is the difference between treatment groups (6g TRC101 QD - Pooled Placebo) in the mean change from baseline = 0 mEq/L; Difference between group LS means = 3.7, 95% CI 2-sided [2.6 to 4.7], Standard Error of Mean 0.5

9. Secondary Outcome: Change From Baseline in Serum Bicarbonate at Day 15 Comparison Between the TRC101 6g QD Dose Group Versus the TRC101 3g BID Dose Group
Description: Serum bicarbonate at Day 15 minus serum bicarbonate at Baseline for the TRC101 6g QD dose group versus that for the TRC101 3g BID dose group
Time Frame: Baseline and Day 15
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Arm/Group | 3g TRC101 BID | 6g TRC101 QD
Number analyzed (Participants) | 25 | 28
mEq/L | 3.0 (0.4) | 3.5 (0.4)
Statistical Analysis 1: Comparison: 3g TRC101 BID vs 6g TRC101 QD; Test type: Other — Two-group test; p = 0.4214, Mixed Models Analysis — The null hypothesis is that the difference between treatment groups (3g TRC101 BID - 6g TRC101 QD) in the mean change from baseline = 0 mEq/L; Difference between group LS means = -0.5, 95% CI 2-sided [-1.6 to 0.7], Standard Error of Mean 0.6

10. Secondary Outcome: Comparison of the Proportion of Subjects in the TRC101 6g QD Dose Group Whose Serum Bicarbonate Values Increased From Baseline to Day 15 by Greater Than or Equal to 2, 3, or 4 mEq/L Versus Placebo
Description: Comparison of the proportion of subjects whose serum bicarbonate values increased from Baseline to Day 15 by greater than or equal to 2, 3, or 4 mEq/L between the 6g TRC101 QD Dose Group versus Placebo
Time Frame: Baseline and Day 15
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | 6g TRC101 QD
Number analyzed (Participants) | 31 | 28
Participants
  => 2 mEq/L Baseline Serum Bicarbonate | 4 | 23
  => 3 mEq/L Baseline Serum Bicarbonate | 2 | 14
  => 4 mEq/L Baseline Serum Bicarbonate | 1 | 12
Statistical Analysis 1: Comparison: Pooled Placebo vs 6g TRC101 QD; Test type: Other — Two-group test; p < 0.0001, Fisher Exact — The null hypothesis is that the difference between treatment groups (6g TRC101 QD - Pooled Placebo) in proportion of subjects whose serum bicarbonate increased from baseline to Day 15 by => 2 mEq/L = 0
Statistical Analysis 2: Comparison: Pooled Placebo vs 6g TRC101 QD; Test type: Other — Two-group test; p = 0.0003, Fisher Exact — The null hypothesis is that the difference between treatment groups (6g TRC101 QD - Pooled Placebo) in the proportion of subjects whose serum bicarbonate increased from baseline to Day 15 by => 3 mEq/L = 0
Statistical Analysis 3: Comparison: Pooled Placebo vs 6g TRC101 QD; Test type: Other — Two-group test; p = 0.0003, Fisher Exact — The null hypothesis is that the difference between treatment groups (6g TRC101 QD - Pooled Placebo) in the proportion of subjects whose serum bicarbonate increased from baseline to Day 15 by => 4 mEq/L = 0

ADVERSE EVENTS:
Time Frame: Through treatment period completion (Day 15)
Description: All subjects completed dosing per protocol and are included in the safety results.
Groups:
- Pooled Placebo: Pooled Placebo treatment group (Placebo administered twice daily [BID] for 14 days + Placebo administered once daily [QD] for 14 days)
Arm/Group | Pooled Placebo | 1.5g TRC101 BID | 3g TRC101 BID | 4.5g TRC101 BID | 6g TRC101 QD
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/25 | 0/25 | 0/26 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/25 | 0/25 | 0/26 | 0/28
Other Adverse Events (participants affected / at risk) | 12/31 | 13/25 | 9/25 | 17/26 | 13/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=31) | 1.5g TRC101 BID (N=25) | 3g TRC101 BID (N=25) | 4.5g TRC101 BID (N=26) | 6g TRC101 QD (N=28)
Diarrhoea (Gastrointestinal disorders) | 4 | 9 | 3 | 6 | 3
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 3
Glomerular filtration rate decreased (Investigations) | 2 | 2 | 1 | 1 | 0
Blood glucose increased (Investigations) | 2 | 1 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 2 | 0
Headache (Nervous system disorders) | 1 | 4 | 1 | 2 | 1
Hypertension (Vascular disorders) | 1 | 1 | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes